CLINICAL TRIAL: NCT03478332
Title: Yangxinshi Pills Plus Conventional Treatment Versus Placebo Plus Conventional Treatment on the Exercise Tolerance of the Patients With Coronary Heart Disease: a Multi-center,Randomised Controlled Clinical Trial
Brief Title: Effects of Yangxinshi Pills on the Exercise Tolerance of the Patients With Coronary Heart Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Changchun University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoping Meng, chief physician, Affiliated Hospital of Changchun University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFH-C04
Record Dates: First submitted 2018-02-11; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Yangxinshi

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): The aim of the arm is to test if the addition of Yangxinshi pills to the conventional coronary heart disease medicine will improve the exercise tolerance of the coronary heart disease
  Interventions: Drug: Yangxinshi pill; Drug: conventional coronary heart disease medicine
- Control group (Placebo Comparator): The patients of the control group are treated with conventional coronary heart disease medicine plus the placebos-Yangxinshi simulant
  Interventions: Drug: conventional coronary heart disease medicine; Drug: Placebos

INTERVENTIONS:
Drug: Yangxinshi pill — 0.6g/tablet
  Other Names: STATE MEDICAL PERMISSION No.Z37021103
  Arms: Treatment group
Drug: conventional coronary heart disease medicine — the conventional treatment includes medicines treating coronary heart disease
  Other Names: glyceryl trinitrate， beta-Blocking agent，etc
Drug: Placebos — Yangxinshi simulant
  Other Names: Yangxinshi simulant
  Arms: Control group

SUMMARY:
Compared with conventional treatment of the coronary heart disease,the aim of the research is to find out if the addition of Yangxinshi pills on the basis of conventional treatment can improve exercise tolerance of patients with coronary heart disease, improve quality of life or restore social function and mental health

DETAILED DESCRIPTION:
90 outpatients with clear diagnosis of coronary heart diseases will be recruited in the trial and randomized into two group.

One group are treated with Yangxinshi pills (provided by Qingdao Growtful Pharmaceutical Co., Ltd.) plus conventional medicine, the other group are treated with placebo plus conventional medicine.

The primary end point is VO2max measured by cardiopulmonary exercise test after 3 months of treatment.

The secondary endpoint is:

1. Mets, Anaerobic threshold（AT）measured by cardiopulmonary exercise test；
2. Changes of other composite indicators of treadmill exercise test or cardiopulmonary exercise test；
3. The maximum walking distance of 6-minute walk test;
4. Changes of Seattle Angina Questionnaire;
5. Hamilton Depression Scale/ Hamilton Anxiety Scale.

The safety evaluation criteria is:

1. Adverse event and serious adverse event;
2. Vital signs;
3. Resting 12 lead ECG;
4. Blood routine examination , urine routine examination、liver and renal function examination(AST、ALT、BUN、Cr).

ELIGIBILITY:
Inclusion Criteria:

* Age 40 ~ 75, gender is not limited
* Have a clear history or ECG of hospital myocardial infarction , diagnosed as coronary heart disease by imaging diagnosis
* Sign the informed consent voluntarily

Exclusion Criteria:

* History of hospitalization for acute coronary syndrome in past 3 months
* Uncontrolled grade 3 hypertension（≥180/100mmHg）or hypotension（<90/60mmHg）
* History of stroke (cerebral hemorrhage, subarachnoid hemorrhage, cerebral thrombosis, cerebral embolism and stroke of unknown type) or lower extremity arterial disease in the past 6 months
* In past 6 months, have medical history of: pregnancy, prepare or suspected of pregnancy, abortion, breastfeeding or after childbirth
* Combined episode bronchial asthma or chronic obstructive pulmonary disease, bradycardia (resting heart rate <60bpm) or atrioventricular block
* Severely allergic constitution, known or likely to be allergic to the test drug or its components
* Known bleeding tendency or hemorrhagic disease
* Patients with severe liver and kidney dysfunction (creatinine clearance ≤ 40ml / min or in the active stage of kidney disease, serum aminotransferase ≥ 2 × upper limit of clinical reference), other life-threatening serious primary or psychiatric diseases and malignant tumors
* Any other situations that researchers believe may affect the clinical research

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05-02 (Estimated); Study Completion 2020-08-25 (Estimated)

PRIMARY OUTCOMES:
change in the maximum volume of O2 consumption | from baseline to 6 months
  measured by gas analyzer

SECONDARY OUTCOMES:
change in exercise tolerance | from baseline to 6 months
  assessed by the distance (in meters) walked on 6-minute walk test
change in left ventricular ejection fraction (in percentage) | from baseline to 6 months
  assessed by echocardiographic examination

OTHER OUTCOMES:
Adverse events | 24 months
  Number of treatment-related adverse events as assessed by CTCAE4.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Meng, Doctor, Principal Investigator — Changchun Traditional Medicine University Affiliated Hospital
Locations (1):
- Changchun Traditional Medicine University Affiliated Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided